CLINICAL TRIAL: NCT01055496
Title: AN OPEN-LABEL, PHASE 1 STUDY OF R-CVP OR R-GDP IN COMBINATION WITH INOTUZUMAB OZOGAMICIN IN SUBJECTS WITH CD22-POSTIVE NON-HODGKIN'S LYMPHOMA
Brief Title: Study Evaluating Chemotherapy in Combination With Inotuzumab Ozogamicin In Subjects With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3129K2-1105; B1931003 (Other: Alias Study Number); 2009-015497-35 (EudraCT Number)
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Lymphoma, B-Cell
Keywords: Non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (R-CVP) (Experimental): Subjects in arm 1 will be enrolled in dose escalation cohorts that will initially evaluate an escalating dose of cyclophosphamide in combination with set doses of inotuzumab ozogamicin, vincristine, prednisone, and rituximab.
  Interventions: Drug: inotuzumab ozogamicin+rituximab +cyclophosphamide+vincristine+prednisone
- Arm 2 (R-GDP) (Experimental): Subjects in arm 2 will be enrolled in dose escalation cohorts that will initially evaluate escalating doses of gemcitabine and/or cisplatinum in combination with set doses of inotuzumab ozogamicin, dexamethasone, and rituximab.
  Interventions: Drug: inotuzumab ozogamicin+rituximab+gemcitabine+cisplatinum+dexamethasone

INTERVENTIONS:
Drug: inotuzumab ozogamicin+rituximab +cyclophosphamide+vincristine+prednisone — Day 1:
  Rituximab at 375 mg/m2 Cyclophosphamide at 375 mg/m2 (cohort 1), 550mg/m2 (cohort 2), 750 mg/m2 (cohort 3, 4) Vincristine at 1.4 mg/m2 (max 2 mg)
  Day 2 Inotuzumab ozogamicin at 0.8 mg/m2 (cohort 1, 2, 3), 1.3 mg/m2 (cohort 4)
  Days 1-5:
  Prednisone at 40 mg/m2
  Each cycle is 3 weeks, with a maximum of 6 cycles total.
  Other Names: CMC-544
  Arms: Arm 1 (R-CVP)
Drug: inotuzumab ozogamicin+rituximab+gemcitabine+cisplatinum+dexamethasone — Day 1:
  Rituximab at 375 mg/m2 Gemcitabine at 500 mg/m2 (cohort 1, 2b, 3b), 1000mg/m2 (cohort 2a, 3a, 4, 5) Cisplatin at 37.5 mg/m2 (cohort 1, 2a), 50mg/m2 (cohort 2b, 3a), 75mg/m2 (cohort 3b, 4, 5)
  Day 2:
  Inotuzumab ozogamicin at 0.8 mg/m2 (cohort 1, 2a, 2b, 3a, 3b, 4), 1.3mg/m2 (cohort 5)
  Days 1-4:
  Dexamethasone at 40 mg
  Each cycle is 3 weeks, with a maximum of 6 cycles total.
  Other Names: CMC-544
  Arms: Arm 2 (R-GDP)

SUMMARY:
This is a phase 1 trial designed to evaluate safety and tolerability of chemotherapy in combination with inotuzumab ozogamicin, an investigational product, in adults with CD22-positive non-Hodgkin's lymphoma. The trial will involve two arms. In one arm, subjects will receive chemotherapy regimen R-CVP (rituximab, cyclophosphamide, vincristine and prednisone). In the other arm, subjects will receive R-GDP (rituximab, gemcitabine, cisplatinum and dexamethasone). Subjects in both arms will also receive inotuzumab ozogamicin.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation cohorts: subjects with diagnosis of CD22-positive Non-Hodgkin's Lymphoma (NHL) who have had at least 1 prior anticancer treatment, including prior treatment with rituximab and chemotherapy.
* Expanded maximum tolerated dose (MTD) confirmation and preliminary efficacy cohorts: subjects with diagnosis of CD22-positive NHL who have had at least 1 prior anticancer treatment, including prior treatment with rituximab and chemotherapy or newly diagnosed subjects who are not candidates for anthracycline-based therapy.
* At least 1 measurable disease lesion that is > 1 cm in the longest transverse diameter, with a product of the diameters > 2.25 cm2 by CT or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Candidate for potentially curative therapy such as stem cell transplantation.
* Prior allogeneic hematopoietic stem cell transplantation (HSCT).
* Prior autologous transplantation, radioimmunotherapy, or other anti CD22 immunotherapy <= 6 months before the first dose of investigational product.
* More than 3 previous combination chemotherapy (2 or more cytotoxics) anticancer regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (10):
  - Davis Cancer Pavillion and Shands Medical Plaza, Gainesville, Florida
  - Shands Cancer Hospital At The University Of Florida, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Gig Harbor, Washington
  - Northwest Medical Specialties, PLLC, Lakewood, Washington
  - Rainier Physicians, PC, Puyallup, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (3):
  - Hopital Saint-Louis -Universite Paris VII, Paris
  - Hospital Saint-Louis - Service d'Hemato-Oncologie, Paris
  - Centre Hospitalier Lyon Sud - Service d'Hematologie, Pierre-Bénite
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Japan (3):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Japanese Foundation For Cancer Research, Koto-Ku, Tokyo
- Singapore General Hospital, Singapore, Singapore
- Samsung Medical Center, Seoul, South Korea
- United Kingdom (4):
  - Nuffield Hospital, Eastleigh, Hants
  - Spire Southampton Hospital, Southampton, Hants
  - Cancer Sciences Division, Somers Cancer Research Building, Southampton, Hants
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sangha R, Davies A, Dang NH, Ogura M, MacDonald DA, Ananthakrishnan R, Paccagnella ML, Vandendries E, Boni J, Goh YT. Phase 1 study of inotuzumab ozogamicin combined with R-GDP for the treatment of patients with relapsed/refractory CD22+ B-cell non-Hodgkin lymphoma. J Drug Assess. 2017 Aug 16;6(1):10-17. doi: 10.1080/21556660.2017.1315336. eCollection 2017. PMID 28959500
- [Derived] Ogura M, Tobinai K, Hatake K, Davies A, Crump M, Ananthakrishnan R, Ishibashi T, Paccagnella ML, Boni J, Vandendries E, MacDonald D. Phase I Study of Inotuzumab Ozogamicin Combined with R-CVP for Relapsed/Refractory CD22+ B-cell Non-Hodgkin Lymphoma. Clin Cancer Res. 2016 Oct 1;22(19):4807-4816. doi: 10.1158/1078-0432.CCR-15-2488. Epub 2016 May 6. PMID 27154915
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K2-1105&StudyName=Study%20Evaluating%20Chemotherapy%20in%20Combination%20With%20Inotuzumab%20Ozogamicin%20In%20Subjects%20With%20Non-Hodgkin%27s%20Lymphoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening included CD-20 & CD-22 immunophenotyping of NHL, international prognostic index or follicular lymphoma international prognostic index score, B-symptom and lymphoma evaluation, Eastern Cooperative Oncology Group performance status, left ventricular ejection fraction assessment, computed tomography scans, bone marrow aspirate and/or biopsy.
Groups:
- Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin: IV inotuzumab ozogamicn (0.8 or 1.3 mg/m^2 on Day 2 of each 21-day cycle) in combination with rituximab (375 mg/m^2) and vincristine (1.4mg/m^2) administererd IV on day 1, prednisone (40mg/m^2) PO on Day 1-5 and cyclophosphamid IV (375, 550 or 750 mg/m^2) on Day 1 of each 21-day cycle (R-CVP) for a maximum of 6 cycles.
- Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin: IV inotuzumab ozogamicin (0.8 mg/m^2 on Day 2 of each 21-day cycle) in combination with IV Rituximab (375 mg/m^2 on Day 1), dexamethasone (40 mg PO on Days 1 to 4), and escalating doses of IV gemcitabine (500 or 1000 mg/m^2) or IV cisplatinum (0, 37.5, 50 or 75 mg/m^2) on Day 1 of each 21-day cycle (R-GDP) for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin
Started | 48 | 55
Completed | 33 | 25
Not Completed | 15 | 30
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 13 | 23
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other - Unspecified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin | Total
Number analyzed (Participants) | 48 | 55 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age measure using mean with Standard deviation
  Years | 62.2 (9.0) | 62.1 (11.8) | 62.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 21 | 18 | 39
    Male | 27 | 37 | 64

OUTCOME MEASURES:

1. Primary Outcome: Participants Reporting Dose Limiting Toxicity (DLT) Adverse Events (AEs) for Participants in the DE Cohort and the MTD Confirmation Cohort for Arm 1
Description: DLT was defined as: febrile neutropenia, Grade (Gr) 4 neutropenia ≥7 days, Gr 4 thrombocytopenia ≥7 days, Gr 3/4 thrombocytopenia associated with bleeding requiring a transfusion, Gr 3/4 non-hematologic toxicity (except alopecia) ≥7 days or treatment-related and clinically significant irrespective of duration, ≥Gr 3 QTc prolongation, Gr 4 alanine or aspartate aminotransferase, Gr 2 hyperbilirubinemia (greater than (>)1.5 x upper normal limit) >7 days, delayed recovery from a treatment-related toxicity that prevented re-dosing by >7 days, or Granulocyte-colony stimulating factor treatment during the first cycle.
Time Frame: From the first dose of study medication (Study Day 1) to the completion of the first 21-day cycle.
Population: Safety Analysis Population includes all subjects who received at least 1 cycle of study drug. Analysis population for DLT is participants evaluable for DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Arm 1: Participants in cohort 1 of Arm 1 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in with combination rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) administered IV on Day 1, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV on Day 1 at a dose of 375 mg/m^2.
- Cohort 2, Arm 1: Participants in cohort 2 of Arm 1 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) administered IV on Day 1, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV on Day 1 at a dose of 550 mg/m^2.
- Cohort 3, Arm 1: Participants in cohort 3 of Arm 1 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) administered IV on Day 1, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV on Day 1 at a dose of 750 mg/m^2.
- Cohort 4, Arm 1: Participants in cohort 4 of Arm 1 received inotuzumab ozogamicin (1.3 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) administered IV on Day 1, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV on Day 1 at a dose of 750 mg/m^2.
- MTD Confirmation Cohort, Arm 1: Participants in the MTD of Arm 1 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) administered IV on Day 1, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV at a dose of 750 mg/m^2.
Arm/Group | Cohort 1, Arm 1 | Cohort 2, Arm 1 | Cohort 3, Arm 1 | Cohort 4, Arm 1 | MTD Confirmation Cohort, Arm 1
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 10
Participants | 0 | 0 | 1 | 2 | 2

2. Secondary Outcome: Percentage of Participants With a Best OR of CR or PR According to International Response Criteria for NHLs in the DE Cohorts
Description: OR was evaluated according to the International Response Criteria for NHLs. CR was defined as complete disappearance of all lesions and disease-related symptoms; all nodes must have decreased to normal (≤1.5 cm in their GTD for nodes >1.5 cm before therapy) or ≤1 cm (short axis) in previously involved node; enlarged spleen prior to therapy must have regressed and be non-palpable; bone marrow lymphoma: infiltrate must have been cleared on repeat bone marrow aspirate and biopsy. PR was defined as >50% decrease in the SPD of up to 6 index lesions. No increase in size of other nodes, liver or spleen. Splenic and hepatic nodules must have regressed by ≥50% in the SPD or GTD (for single nodules). With the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. No progression of non-target disease or new lesions.
Time Frame: From first dose of study medication through 2 year follow-up period, including but not limited to planned assessments scheduled every 9 to 24 weeks.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- DE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin: Participants received inotuzumab ozogamicin (0.8 or 1.3 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with R-CVP. Rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) were administered IV on Day 1, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV at escalating doses of 375, 550, or 750 mg/m^2 on Day 1, of each 21-day cycle for a maximum of 6 cycles, according to a 3+3 DE rule where the doses escalated in a step-by-step fashion to determine the MTD.
- DE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin: Participants received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with R-GDP. Rituximab (375 mg/m^2) was administered IV on Day 1 and dexamethasone (40 mg) PO on Days 1 to 4. Participants received escalating doses of gemcitabine (500 or 1000 mg/m^2) or cisplatinum (0, 37.5, 50 or 75 mg/m^2) and were administered IV on Day 1 of each 21-day cycle, for a maximum of 6 cycles. DE in Arm 2 was conducted using an up-and-down dose escalation method by increasing or decreasing the dose of either cisplatinum or gemcitabine to determine the MTD.
Arm/Group | DE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | DE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 16 | 27
Percentage of participants | 81.3 [54.35 to 95.95] | 51.9 [31.95 to 71.33]

3. Primary Outcome: Participants Reporting DLT AEs for Participants in the DE Cohort and the MTD Confirmation Cohort for Arm 2
Description: as for outcome 1
Time Frame: From the first dose of study medication (Study Day 1) to the completion of the first 21-day cycle.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1, Arm 2: Participants in cohort 1 of Arm 2 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and gemcitabine (500 mg/m^2) and cisplatinum (37.5 mg/m^2) administered IV on Day 1 of each 21-day cycle.
- Cohort 2a, Arm 2: Participants in cohort 2a of Arm 2 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and gemcitabine (1000 mg/m^2) and cisplatinum (37.5 mg/m^2) administered IV on Day 1 of each 21-day cycle.
- Cohort 2b, Arm 2: Participants in cohort 2b of Arm 2 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and gemcitabine (500 mg/m^2) and cisplatinum (50 mg/m^2) administered IV on Day 1 of each 21-day cycle.
- Cohort 3b, Arm 2: Participants in cohort 3b of Arm 2 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and gemcitabine (500 mg/m^2) and cisplatinum (75 mg/m^2) administered IV on Day 1 of each 21-day cycle.
- Cohort 4, Arm 2: Participants in cohort 4 of Arm 2 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and gemcitabine (1000 mg/m^2) administered IV on Day 1 of each 21-day cycle.
- MTD Confirmation Cohort, Arm 2: Participants in the MTD cohort of Arm 2 received inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles in combination with rituximab (375 mg/m^2), cisplatinum (50 mg/m^2) and gemcitabine (500 mg/m^2) IV on Day 1, and dexamethasone (40 mg) PO on Days 1 to 4 of each 21-day cycle.
Arm/Group | Cohort 1, Arm 2 | Cohort 2a, Arm 2 | Cohort 2b, Arm 2 | Cohort 3b, Arm 2 | Cohort 4, Arm 2 | MTD Confirmation Cohort, Arm 2
Number analyzed (Participants) | 6 | 3 | 8 | 4 | 6 | 10
Participants | 0 | 2 | 1 | 2 | 0 | 3

4. Primary Outcome: Percentage of Participants With Best Overall Response (OR) of Complete Response (CR) or Partial Response (PR) According to International Response Criteria for NHLs in the MTD and EE Cohorts
Description: OR was evaluated according to the International Response Criteria for NHLs. CR was defined as complete disappearance of all lesions and disease-related symptoms; all nodes must have decreased to normal (less than or equal to [≤]1.5 centimeters [cm] in their greatest transverse diameter (GTD) for nodes >1.5 cm before therapy) or ≤1 cm (short axis) in previously involved node; enlarged spleen prior to therapy must have regressed and be non-palpable; bone marrow lymphoma: infiltrate must have been cleared on repeat bone marrow aspirate and biopsy. PR was defined as >50% decrease in the sum of the product diameters (SPD) of up to 6 index lesions. No increase in size of other nodes, liver or spleen. Splenic and hepatic nodules must have regressed by ≥50% in the SPD or GTD (for single nodules). With the exception of splenic and hepatic nodules, involvement of other organs is usually assessable and no measurable disease should be present. No progression of non-target disease or new lesions.
Time Frame: as for outcome 2
Population: Intent-to-Treat (ITT) population: all participants enrolled into the study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin: Participants received rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) IV on Day 1, inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 and prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV at 750 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 6 cycles.
- MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin: Participants received rituximab (375 mg/m^2), cisplatinum (50 mg/m^2) and gemcitabine (500 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles.
Arm/Group | MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 32 | 28
Percentage of participants | 81.3 [63.56 to 92.79] | 53.6 [33.87 to 72.49]

5. Secondary Outcome: Kaplan-Meier Estimate of the Progression-Free Survival (PFS) in the DE Cohorts
Description: PFS was defined as time from date of first dose to the earlier date of progression (including symptomatic deterioration), date of death from any cause, or initiation of new anticancer therapy for the lymphoma. Participants without an event were censored at the date of the last valid tumour assessment. A valid tumour assessment visit was defined as the tumour assessment visit with overall response of CR, PR, stable disease (SD), or disease progression (PD), but not 'Not Done' or 'Unknown'. Participants without a post-baseline tumour assessment and without a PFS event were censored on the date of first dose.
Time Frame: as for outcome 2
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | DE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 16 | 27
Months | 16.36 [4.40 to 23.39] | 10.12 [3.45 to 28.16]

6. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Alive and Free From PD or New Anticancer Therapy at 6, 12, and 24 Months in the DE Cohorts
Description: Measure includes death from any cause, PD (including symptomatic deterioration) during and after treatment or initiation of new anticancer therapy for the lymphoma. PD was defined as symptomatic deterioration and according to the International Response Criteria for NHL: 1) appearance of any new lesion >1.5 cm in any axis during or at EOT, even if other lesions are decreasing, 2) at least a 50% increase from nadir in the SPD of any previously involved or single involved nodes, or the size of other lesions (splenic or hepatic). Lymph nodes with a short axis diameter of <1.0 cm must increase by ≥50% and to a size of 1.5x1.5 cm or >1.5 cm in the long axis, 3) 50% increase in the longest diameter of any single previously identified node >1 cm in its short axis. PD was defined as clinical PD, new non-nodal lesions or new nodal lesion ≥1.5 cm in GTD, progression of existing non-index lesions or bone marrow that was negative and now positive.
Time Frame: 6, 12 and 24 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | DE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | DE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 16 | 27
Percent Probability
  6 months | 80.00 [49.98 to 93.07] | 60.98 [39.42 to 76.89]
  12 months | 66.67 [37.53 to 84.56] | 47.92 [27.41 to 65.82]
  24 months | 22.22 [4.64 to 47.87] | 33.54 [15.58 to 52.63]

7. Secondary Outcome: Kaplan-Meier Estimate of the PFS in the MTD Confirmation/EE Cohorts
Description: PFS was defined as time from date of first dose to the earlier date of progression (including symptomatic deterioration), date of death from any cause, or initiation of new anticancer therapy for the lymphoma. Participants without an event were censored at the date of the last valid tumour assessment. A valid tumour assessment visit was defined as the tumour assessment visit with OR of CR, PR, SD, or PD, but not 'Not Done' or 'Unknown'. Participants without a post-baseline tumour assessment and without a PFS event were censored on the date of first dose.
Time Frame: as for outcome 2
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 32 | 28
Months | 14.36 [5.13 to NA] — NA means upper limit for 95% CI could not be estimated due to insufficient events observed. | 6.14 [4.44 to 10.64]

8. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Alive and Free From PD or New Anticancer Therapy at 6, 12, and 24 Months in the MTD Confirmation/EE Cohorts.
Description: as for outcome 6
Time Frame: 6, 12, and 24 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 32 | 28
Percent Probability
  6 months | 61.85 [42.66 to 76.26] | 54.74 [31.90 to 72.77]
  12 months | 51.54 [32.83 to 67.41] | 24.88 [9.15 to 44.52]
  24 months | 44.67 [26.73 to 61.12] | NA [NA to NA] — NA means the corresponding parameters could not be estimated due to insufficient events observed.

9. Secondary Outcome: Kaplan-Meier Estimate of the Overall Survival (OS) in the DE Cohorts
Description: OS was defined from date of first dose to date of death due to any cause, censoring at the date of last contact.
Time Frame: From first dose of study medication through 2 year follow-up period
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | DE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | DE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 16 | 27
Months | NA [11.70 to NA] — NA means the corresponding parameters could not be estimated due to insufficient events observed. | NA [7.03 to NA] — NA means the corresponding parameters could not be estimated due to insufficient events observed.

10. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Alive at 6, 12, and 24 Months in the DE Cohorts
Description: OS was defined from date of first dose to date of death due to any cause, censoring at the date of last contact.
Time Frame: 6, 12, and 24 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | DE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | DE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 16 | 27
Percent Probability
  6 months | 100.00 [100.00 to 100.00] | 74.07 [53.19 to 86.70]
  12 months | 80.00 [49.98 to 93.07] | 62.96 [42.12 to 78.07]
  24 months | 80.00 [49.98 to 93.07] | 55.09 [34.62 to 71.53]

11. Secondary Outcome: Kaplan-Meier Estimate of the OS in the MTD Confirmation/EE Cohorts
Description: OS was defined from date of first dose to date of death due to any cause, censoring at the date of last contact.
Time Frame: From first dose of study medication through 2 year follow-up period
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 32 | 28
Months | NA [24.51 to NA] — NA means the corresponding parameters could not be estimated due to insufficient events observed. | NA [8.38 to NA] — NA means the corresponding parameters could not be estimated due to insufficient events observed.

12. Secondary Outcome: Kaplan-Meier Estimates of the Probability of Being Alive at 6, 12, and 24 Months in the MTD Confirmation/EE Cohorts
Description: OS was defined from date of first dose to date of death due to any cause, censoring at the date of last contact.
Time Frame: 6, 12, and 24 Months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 32 | 28
Percent Probability
  6 months | 84.38 [66.46 to 93.18] | 88.00 [67.26 to 95.96]
  12 months | 78.13 [59.52 to 88.92] | 59.11 [37.29 to 75.56]
  24 months | 71.61 [52.51 to 84.11] | 53.74 [31.82 to 71.40]

13. Primary Outcome: Percentage of Participants With a Treatment Emergent AE
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event may not necessarily have had a causal relationship with the treatment or usage. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were defined as those occurring on or after the first study drug dose day through and including 56 days post last dose of study drug. The severity of all AEs was graded by the investigator using the National Cancer Institute Common Terminology Criteria for AE Version 3.0 (NCI CTCAE v3.0).
Time Frame: SAEs were assessed from informed consent through and including the end of treatment visit (at least 28 calendar days after last study drug administration). Non-SAEs were recorded from time of the first dose of study drug through last participant visit.
Population: Safety population - included all participants who received ≥1 cycle of investigational product
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 48 | 55
Percentage of Participants
  Subjects with AEs | 100 | 100
  Subjects with SAEs | 31.3 | 45.5
  Subjects with Grade 3 or 4 AEs | 89.6 | 96.4
  Subjects with Grade 5 AEs | 4.2 | 5.5
  Subjects discontinued due to AEs | 27.1 | 36.4
  Subjects with dose reduced due to AEs | 16.7 | 32.7
  Subjects with temporary discontinuation due to AEs | 54.2 | 67.3

14. Primary Outcome: Percentage of Participants With Any Grade 3/4 Chemistry Abnormality During Therapy
Description: The following parameters were analyzed for blood chemistry: blood urea nitrogen (or urea), creatinine, glucose, calcium, sodium, potassium, phosphorus, lactate dehydrogenase, aspartate aminotransferase, alanine aminotransferase, total bilirubin (and direct bilirubin, if total bilirubin was elevated), alkaline phosphatase, uric acid (or urate), albumin and total protein. Laboratory test results were graded using the NCI CTCAE v3.0 where CTCAE Grade 3 equals "severe" and CTCAE Grade 4 equals "life threatening or disabling."
Time Frame: Within 3 days prior to the start of each cycle, on Day 8 of each cycle, on Day 15 of Cycles 1, 2, and 3, and the end-of-treatment visit. Each Cycle is 21 Days.
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 48 | 55
Percentage of Participants | 21.3 | 36.4

15. Primary Outcome: Percentage of Participants With Any Grade 3/4 Hematology Abnormality During Therapy
Description: The following parameters were analyzed for hematology: lymphocytes, basophils, eosinophils, erythrocytes, hematocrit, hemoglobin, leukocytes, monocytes, neutrophils, platelets, prothrombin international normalized ratio, prothrombin time, fibrinogen, and activated partial thromboplastin time. Laboratory test results were graded using the NCI CTCAE v3.0 where CTCAE Grade 3 equals "severe" and CTCAE Grade 4 equals "life threatening or disabling."
Time Frame: Within 3 days prior to the start of each cycle, Day 8 of each cycle, Day 15 of Cycles 1, 2, and 3, and the end-of-treatment visit. Each Cycle is 21 Days.
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 48 | 55
Percentage of Participants | 91.7 | 96.4

16. Secondary Outcome: Mean Inotuzumab Ozogamicin Serum Concentrations
Description: Pharmacokinetic (PK) samples were required for participants enrolled in the confirmatory and preliminary efficacy MTD cohorts only (Parts 2 and 3). Concentrations of inotuzumab ozogamicin in serum were determined using appropriate, validated unconjugated (also known as free) bioanalytical assays.
Time Frame: Pre-dose on Cycle 1, Day 2; Pre-dose, 1 and 3 hours post-dose on Cycle 3, Day 2; 24 hours post-dose on Cycle 3, Day 3 and 168 hours post-dose on Cycle 3, Day 8.
Population: PK population - included all participants who provided samples for PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 3/MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin: Participants received rituximab (375 mg/m^2) and vincristine (1.4 mg/m^2) IV on Day 1, inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2, prednisone (40 mg/m^2) PO on Days 1 to 5 and cyclophosphamide IV at 750 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 6 cycles.
- Cohort 2b/MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin: Participants received rituximab (375 mg/m^2), cisplatinum (50 mg/m^2) and gemcitabine (500 mg/m^2) IV on Day 1, dexamethasone (40 mg) PO on Days 1 to 4, and inotuzumab ozogamicin (0.8 mg/m^2) IV on Day 2 of each 21-day cycle for a maximum of 6 cycles.
Arm/Group | Cohort 4, Arm 1 | Cohort 1, Arm 2 | Cohort 3b, Arm 2 | Cohort 4, Arm 2 | Cohort 3/MTD/EE Arm 1: (R-CVP) Plus Inotuzumab Ozogamicin | Cohort 2b/MTD/EE Arm 2: (R-GDP) Plus Inotuzumab Ozogamicin
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 38 | 36
ng/mL
  Cycle 1 Day 2, 0h: number analyzed (Participants) | 1 | 3 | 1 | 1 | 31 | 30
  Cycle 1 Day 2, 0h | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0.
  Cycle 3 Day 2, 0h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 23 | 19
  Cycle 3 Day 2, 0h |  |  |  |  | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | 25.00 (76.151)
  Cycle 3 Day 2, 1h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 15
  Cycle 3 Day 2, 1h |  |  |  |  | 189.74 (81.528) | 283.27 (127.151)
  Cycle 3 Day 2, 3h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 15
  Cycle 3 Day 2, 3h |  |  |  |  | 213.95 (71.692) | 280.33 (119.12)
  Cycle 3 Day 3, 24h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 22 | 15
  Cycle 3 Day 3, 24h |  |  |  |  | 110.39 (37.468) | 154.25 (81.608)
  Cycle 3 Day 8, 168h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 19 | 18
  Cycle 3 Day 8, 168h |  |  |  |  | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0. | NA (NA) — Summary statistics are not presented as number of observations above lower limit of quantification (NALQ) = 0.

ADVERSE EVENTS:
Time Frame: SAEs were assessed from informed consent through and including the end of treatment visit (at least 28 calendar days after last study drug administration). Non-SAEs were recorded from time of the first dose of study drug through last participant visit.
Description: Presented SAEs & AEs are treatment-emergent events (occurring on or after first study drug dose through and including 56 days post last dose of study drug).
Arm/Group | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin
Serious Adverse Events (participants affected / at risk) | 15/48 | 25/55
Other Adverse Events (participants affected / at risk) | 48/48 | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin (N=48) | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Device occlusion (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Corynebacterium infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 1 | 3
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (R-CVP) Plus Inotuzumab Ozogamicin (N=48) | Arm 2 (R-GDP) Plus Inotuzumab Ozogamicin (N=55)
Anaemia (Blood and lymphatic system disorders) | 12 | 24
Leukopenia (Blood and lymphatic system disorders) | 31 | 15
Lymphopenia (Blood and lymphatic system disorders) | 28 | 17
Neutropenia (Blood and lymphatic system disorders) | 36 | 38
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 46
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Flushing (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 2 | 4
Abdominal discomfort (Gastrointestinal disorders) | 5 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6
Ascites (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 29 | 24
Diarrhoea (Gastrointestinal disorders) | 8 | 12
Dry mouth (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 4
Haemorrhoids (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 21 | 25
Stomatitis (Gastrointestinal disorders) | 5 | 8
Vomiting (Gastrointestinal disorders) | 10 | 13
Asthenia (General disorders) | 4 | 6
Chest pain (General disorders) | 3 | 0
Chills (General disorders) | 2 | 9
Fatigue (General disorders) | 24 | 29
Malaise (General disorders) | 9 | 1
Mucosal inflammation (General disorders) | 1 | 3
Oedema (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 4 | 11
Pyrexia (General disorders) | 9 | 16
Tachycardia (Cardiac disorders) | 2 | 3
Drug hypersensitivity (Immune system disorders) | 5 | 0
Hypersensitivity (Immune system disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 1
Oral candidiasis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 8
Urinary tract infection (Infections and infestations) | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 4
Fall (Injury, poisoning and procedural complications) | 4 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 2
Alanine aminotransferase increased (Investigations) | 17 | 5
Aspartate aminotransferase increased (Investigations) | 21 | 11
Blood alkaline phosphatase increased (Investigations) | 13 | 6
Blood lactate dehydrogenase increased (Investigations) | 8 | 2
C-reactive protein increased (Investigations) | 4 | 2
Electrocardiogram QT prolonged (Investigations) | 5 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Protein total decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 3 | 5
Haematuria (Renal and urinary disorders) | 3 | 3
Pollakiuria (Renal and urinary disorders) | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 18 | 5
Liver disorder (Hepatobiliary disorders) | 10 | 4
Decreased appetite (Metabolism and nutrition disorders) | 15 | 15
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Dizziness (Nervous system disorders) | 3 | 3
Dysgeusia (Nervous system disorders) | 9 | 7
Headache (Nervous system disorders) | 7 | 5
Hypoaesthesia (Nervous system disorders) | 10 | 1
Neuropathy peripheral (Nervous system disorders) | 11 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2
Agitation (Psychiatric disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 3 | 3
Confusional state (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 12 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 5 | 6

LIMITATIONS AND CAVEATS:
This is a preliminary study with a limited number of participants, which was performed primarily to assess safety.The sample size for this study was determined by clinical rather than statistical considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days